CLINICAL TRIAL: NCT07241325
Title: A Cross-Sectional Observational Study to Evaluate Psychological Well-Being, Depression, and Health-Related Quality of Life and Their Demographic and Clinical Correlates in Adults With Type 2 Diabetes Attending an Outpatient Metabolic Clinic
Brief Title: Psychological Well-Being, Depression, and Health-Related Quality of Life in Adults With Type 2 Diabetes: A Cross-Sectional Study
Acronym: PWDQ-T2D
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202508155RIND
Record Dates: First submitted 2025-09-24; First posted 2025-11-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Health-related Quality of Life; Depressive Symptoms; Psychological Well-being; Spiritual Well-being
Keywords: Type 2 Diabetes Mellitus; Psychological Well-Being; Depression; PHQ-9; EQ-5D-5L; Shalom Scale; Spiritual Well-Being; Psychosocial Support; Cross-Sectional; Observational; Taiwan
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression; Psychological Well-Being

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cross-sectional observational study aims to explore the relationships among psychological well-being, depression, and quality of life in patients with type 2 diabetes attending the outpatient metabolic clinic at National Taiwan University Hospital. The study will collect data using standardized instruments, including the EQ-5D Health-Related Quality of Life Questionnaire, the PHQ-9 Depression Scale, and the Shalom Scale of Psychological Well-Being, along with demographic and clinical variables such as age, sex, education, body mass index, HbA1c, disease duration, and psychosocial support indicators. Descriptive statistics, Pearson correlation analyses, ANOVA, and multiple linear regression modeling will be performed to identify factors associated with psychological well-being. The findings are expected to provide evidence-based insights to inform tailored interventions and improve the mental health and quality of life of patients with type 2 diabetes.

DETAILED DESCRIPTION:
This is a prospective, cross-sectional observational study designed to examine the relationships among psychological well-being, depression, and quality of life in adult patients with type 2 diabetes attending the outpatient metabolic clinic at National Taiwan University Hospital. The study seeks to identify demographic, clinical, and psychosocial factors associated with psychological well-being in this population.

Eligible participants will be ≥18 years old, diagnosed with type 2 diabetes, able to complete self-administered Chinese questionnaires, and willing to provide written informed consent. Patients with major psychiatric disorders, moderate to severe cognitive impairment, acute diabetic complications, or significant communication barriers will be excluded.

Data collection will include demographic variables (e.g., age, sex, education, marital status, religious belief, economic status, family support, sleep quality, exercise habits) and clinical indicators (e.g., diabetes duration, BMI, HbA1c, diabetic complications, estimated glomerular filtration rate). Three standardized instruments will be administered:

EQ-5D-5L to measure health-related quality of life

PHQ-9 to assess depressive symptoms

Shalom Scale to evaluate psychological well-being

The planned sample size is 350 participants. Recruitment will be conducted by the research team during clinic hours. Written informed consent will be obtained before any data collection.

Statistical analyses will include descriptive statistics to summarize participant characteristics and scale scores, Pearson correlation analyses to examine associations between variables, one-way ANOVA to compare psychological well-being across subgroups, and multiple linear regression modeling to identify predictors of psychological well-being.

The study period is from September 2025 to December 2026. This research is investigator-initiated and self-funded. The results will provide an evidence-based foundation for designing tailored clinical and psychosocial interventions to improve mental health and quality of life in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older with full legal capacity.
2. Clinically diagnosed with Type 2 Diabetes Mellitus and receiving ongoing outpatient care.
3. Able to read and understand Chinese questionnaires and complete self-administered forms.
4. Understand the study purpose and procedures and provide written informed consent.

Exclusion Criteria:

1. Presence of major psychiatric disorders (e.g., schizophrenia, bipolar disorder, major depressive disorder).
2. Moderate to severe cognitive impairment or dementia, as assessed by the clinical physician, making it impossible to complete the questionnaires.
3. Currently experiencing acute diabetic complications (e.g., diabetic ketoacidosis, hyperosmolar hyperglycemic state) or hospitalization.
4. Severe language or other communication barriers preventing expression of consent or understanding of study content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (aged 18 years and older) with a confirmed diagnosis of type 2 diabetes mellitus receiving ongoing outpatient care at the Metabolism Clinic of National Taiwan University Hospital. Approximately 350 participants will be recruited using convenience sampling during routine clinic visits. All participants must be able to read and understand Chinese questionnaires, complete self-administered forms, and provide written informed consent. The study does not include healthy volunteers or individuals without type 2 diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Shalom Scale Total Score (Psychological Well-Being) | At enrollment (single outpatient visit; questionnaires completed in approximately 30-40 minutes).
  The Shalom Scale for Psychological Well-Being will be used to measure psychological well-being. Higher scores indicate better spiritual/psychological well-being. The total score will be analyzed as a continuous variable.

SECONDARY OUTCOMES:
PHQ-9 Total Score (Depression Severity) | Day 1
  The Patient Health Questionnaire-9 (PHQ-9) will be used to assess the severity of depressive symptoms. Total scores range from 0 to 27, where higher scores indicate more severe depression.
EQ-5D-5L Index Score (Health Utility) | Day 1
  The EQ-5D-5L index score will be used to assess health-related quality of life using the Taiwan value set. Index scores typically range from below 0 (health states worse than death) to 1.0 (full health), with higher scores indicating better health status.
EQ-5D-5L Visual Analog Scale (VAS) | Day 1
  The EQ-5D-5L Visual Analog Scale (VAS) will be used to assess patients' self-rated overall health status. Scores range from 0 (worst imaginable health) to 100 (best imaginable health), with higher scores indicating better perceived health.

OTHER OUTCOMES:
Associations Between Demographic/Clinical Variables and Psychological Well-Being | Day 1
  Associations between psychological well-being and demographic or clinical variables will be examined using correlation and multivariable regression analyses. Pearson correlation (r) will be used to assess bivariate associations between the Shalom Scale total score and PHQ-9 total score, EQ-5D-5L index score, and HbA1c (%). Multiple linear regression analyses will be performed to estimate standardized beta coefficients (β) for predictors of Shalom Scale total score, including age, sex, diabetes duration, BMI, HbA1c, presence of complications, family support, sleep quality, and exercise frequency. Results will be reported as correlation coefficients (r) or standardized β coefficients (unitless).
Exploratory Subgroup Analyses of Psychological Well-Being, Depression, and Quality of Life | Day 1
  Exploratory subgroup analyses will be conducted to examine differences in psychological well-being, depression severity, and health-related quality of life across demographic or clinical subgroups. Subgroups of interest include sex (male vs. female), age group (e.g., <65 vs. ≥65 years), diabetes duration (short vs. long duration), and presence of diabetes-related complications. Group comparisons will be performed using t-tests or ANOVA as appropriate. Results will be reported as mean differences in scores between subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yuan Wang, Principal Investigator — National Taiwan University Hospital, Department of Internal Medicine (Metabolism)
Locations (1):
- National Taiwan University Hospital - Metabolism, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that may be shared include questionnaire scores and coded demographic and clinical variables (e.g., age group, sex, diabetes duration, BMI category, HbA1c range, presence of complications). No directly identifiable information (such as names, ID numbers, or contact information) will be included. Data will be stored and shared only under institutional data-sharing agreements, following approval by the National Taiwan University Hospital Research Ethics Committee.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 12 months after publication of the main results; available for up to 5 years thereafter.
Access Criteria: Qualified researchers may request access by submitting a written proposal and institutional data-sharing agreement to the Principal Investigator. Approval will be required from the National Taiwan University Hospital Research Ethics Committee prior to data release.
URL: https://www.ntuh.gov.tw/RE/

REFERENCES:
- [Result] Shalom S., Wang Y.T., Wang C.H., Hu R.Z. (2013). Development and validation of the Shalom Scale for psychological well-being in Chinese populations. Fu Jen Medical Journal, 11(3), 197-204.
- [Result] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941

DOCUMENTS (2):
  • Study Protocol (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT07241325/Prot_000.pdf
  • Informed Consent Form (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT07241325/ICF_001.pdf